CLINICAL TRIAL: NCT04638309
Title: Phase 1 Study to Evaluate Safety and Efficacy of APR-548 in Combination With Azacitidine for the Treatment of TP53-Mutant Myelodysplastic Syndromes
Brief Title: APR-548 in Combination With Azacitidine for the Treatment of TP53 Myelodysplastic Syndromes (MDS)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Aprea Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A20-11202
Record Dates: First submitted 2020-11-13; First posted 2020-11-20 (Actual); Results first posted 2025-03-07 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: MDS; Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Dose level 1
  Interventions: Drug: APR-548 + Azacitidine
- Cohort 2 (Experimental): Dose level 2
  Interventions: Drug: APR-548 + Azacitidine
- Cohort 3 (Experimental): Dose level 3
  Interventions: Drug: APR-548 + Azacitidine

INTERVENTIONS:
Drug: APR-548 + Azacitidine — APR-548 monotherapy period followed by APR-548 in combination with Azacitidine

SUMMARY:
Phase 1 study evaluating the safety and efficacy of APR-548 in combination with Azacitidine for the treatment of TP53-Mutant Myelodysplastic Syndromes.

DETAILED DESCRIPTION:
Open-label first-in-human (FIH) phase 1 clinical trial assessing the safety, pharmacokinetics (PK), and clinical activity of orally (p.o.) administered APR-548 alone and in combination with azacitidine for the treatment of TP53-mutant myelodysplastic syndromes (MDS).

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent prior to any study specific procedures.
2. Documented diagnosis of TP53-mutant MDS, according to WHO criteria that is relapsed/refractory or previously untreated MDS.
3. Adequate organ function as defined by the following laboratory values:

   1. Creatinine clearance ≥60 mL/min (by Cockcroft-Gault method, Appendix I),
   2. Total serum bilirubin ≤1.5 × upper limit of normal (ULN) unless due to Gilbert's syndrome or MDS organ involvement,
   3. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 × ULN, unless due to MDS organ involvement.
4. Age ≥18 years at the time of signing the informed consent form.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2 (Appendix II).
6. Projected life expectancy of ≥12 weeks.
7. Clear ocular media and adequate pupil dilation to permit fundus examination and retinal imaging.

Exclusion Criteria:

1. Cardiac abnormalities, which includes, but not limited to:

   1. Myocardial infarction within six months prior to enrollment
   2. New York Heart Association Class III or IV heart failure or known LVEF <40%
2. Concomitant malignancies or previous malignancies with less than a 1 year disease-free interval at the time of signing informed consent.
3. Use of cytotoxic chemotherapeutic agents, or experimental agents for the treatment of MDS within 14 days or 5 half-lives of the product (whichever is shorter) of the first day of study drug treatment.
4. Prior exposure to eprenetapopt (APR-246).
5. A female subject who is pregnant or breast-feeding.
6. Known history of human immunodeficiency virus (HIV), active hepatitis B or active hepatitis C infection.
7. Malabsorption syndrome or other condition likely to affect gastrointestinal absorption of APR-548.
8. Known history or current evidence of ocular disease in either eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Gullbo, MD, Study Director — Theradex Oncology
Locations (4):
- United States (4):
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institue, Boston, Massachusetts
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was terminated prior to enrollment into cohort 2 and 3.
Groups:
- Cohort 1: Dose level 1
  APR-548 50 mg/d + Azacitidine 75 mg/d: APR-548 monotherapy period followed by APR-548 in combination with Azacitidine
- Cohort 2: Dose level 2
  APR-548 150 mg/d + Azacitidine 75 mg/d: APR-548 monotherapy period followed by APR-548 in combination with Azacitidine
- Cohort 3: Dose level 3
  APR-548 300 mg/d + Azacitidine 75 mg/d: APR-548 monotherapy period followed by APR-548 in combination with Azacitidine
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Started | 4 | 0 | 0
Completed | 3 | 0 | 0
Not Completed | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study was terminated.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Total
Number analyzed (Participants) | 4 | 0 | 0 | 4
Age, Continuous [Median (Full Range); unit: years] | 64 [58 to 74] |  |  | 64 [58 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 0 | 3
  Male | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  |  | 0
  Asian | 0 |  |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  |  | 0
  Black or African American | 0 |  |  | 0
  White | 4 |  |  | 4
  More than one race | 0 |  |  | 0
  Unknown or Not Reported | 0 |  |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 |  |  | 4

OUTCOME MEASURES:

1. Primary Outcome: To Investigate the "Number of Participants With Treatment Emergent Adverse Events From Treatment With APR-548 as Monotherapy and in Combination With Azacitidine
Description: Occurrence of frequency of treatment emergent adverse events by reviewing safety data including AEs, vital signs, laboratory data, ECG, ophthalmologic assessment findings, and other physical exam findings.
Time Frame: Through study completion, approximately 28 days
Population: Study was terminated.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1
Number analyzed (Participants) | 3
Participants | 3

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Cohort 1
All-Cause Mortality (participants affected / at risk) | 2/4
Serious Adverse Events (participants affected / at risk) | 2/4
Other Adverse Events (participants affected / at risk) | 2/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=4)
Fall (Injury, poisoning and procedural complications) | 1
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Sinusitis (Infections and infestations) | 1
Stroke (Vascular disorders) | 1 (2)
Myocardial Infarcation (Cardiac disorders) | 1
Cardiogenic Shock (Cardiac disorders) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=4)
Alkaline phosphatase increase (Investigations) | 1
Drug hypersensitivity (General disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Candida Infection (Infections and infestations) | 1
Confusional state (Psychiatric disorders) | 1
Contusion (Injury, poisoning and procedural complications) | 2
Dehydration (General disorders) | 1
Depression (Psychiatric disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2 (4)
Dizziness (General disorders) | 1
Dysphemia (Psychiatric disorders) | 1
Extrapyramidal disorder (Nervous system disorders) | 1
Fatigue (General disorders) | 2
Flatulence (Gastrointestinal disorders) | 1
Flushing (Skin and subcutaneous tissue disorders) | 1
hemorrhoids hemmorage (General disorders) | 1
Headache (General disorders) | 1 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypersomnia (Psychiatric disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Infusion site pruritis (Skin and subcutaneous tissue disorders) | 1
Ingrown Nail (Skin and subcutaneous tissue disorders) | 1
Lactic Acidosis (Metabolism and nutrition disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Odema Peripheral (Vascular disorders) | 1 (3)
Pain in extremity (General disorders) | 1
Periorbital Edema (Eye disorders) | 1
Phlebitis (Vascular disorders) | 1
Tremor (Nervous system disorders) | 1
urinary hestiation (Renal and urinary disorders) | 1
Vison Blurred (Eye disorders) | 1
Vision Impairment (Eye disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-10): https://cdn.clinicaltrials.gov/large-docs/09/NCT04638309/Prot_SAP_000.pdf